CLINICAL TRIAL: NCT00756899
Title: The Relationship Between Vitamin D Deficiency and Low Bone Mineral Content in Children
Brief Title: Vitamin D Deficiency and Low Bone Mineral Content in Children
Acronym: VDS
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Benjamin U. Nwosu, Study Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: H-12795
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Vitamin D Deficiency; Obesity
Keywords: Vitamin D deficiency, insulin resistance, obesity, bone
MeSH Terms: conditions — Vitamin D Deficiency; Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Obese: Chilren with BMI of >95th percentile
- Non-obese: Children with BMI of <85th percentile

SUMMARY:
The Vitamin D study is designed to investigate the effect of body fat mass on vitamin D levels in children. Earlier studies have shown that individuals with increased fat mass may have low vitamin D levels.

Our specific hypothesis states that children with increased fat mass will have lower blood levels of vitamin D when compared to non-obese children.Since vitamin D is the primary hormone for bone mineralization in humans, low levels of vitamin D could lead to decreased bone mineral content in these children.

DETAILED DESCRIPTION:
Fifty prepubertal male and female children of ages between 3-12 years will participate in this study. Of these, 25 obese children will be enrolled in the study group, and 25 non-obese children will serve as controls.

All subjects will fill out a comprehensive mineral intake questionnaire as part of the study to ensure adequate calcium intake prior to the study.

All subjects will collect a first morning urine sample for calcium, creatinine, and NTX.

Fasting blood samples will be drawn for the following analytes: 25-hydroxyvitamin D, 1, 25-dihydroxyvitamin D, intact PTH, calcium, phosphorus, magnesium, osteocalcin, insulin, c-peptide, fasting blood glucose, leptin, and adiponectin.

Bone Mineral Content will be evaluated in 16 obese subjects with vitamin D level of < 30 nmol/L.

ELIGIBILITY:
Inclusion Criteria:

* General: Prepubertal children (males, with testicular volume of ≤ 3 cc, and girls with Tanner 1 breast) of ages 7-11 years will be enrolled in the study.
* Study group: Subjects with a BMI of > 95th percentile for age and sex.
* Control group: All control subjects will have a BMI of < 85th percentile for age and sex.

Exclusion Criteria:

* known metabolic or genetic diseases resulting in obesity such as severe hypothyroidism, pseudohypoparathyroidism, or Cushing's disease
* diabetes mellitus
* subjects on lipid lowering medications
* subjects on medications known to impact body weight or calcium homeostasis
* subjects with a history of recent significant weight loss or gain

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Prepubertal children
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Bone mineral content | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin U Nwosu, MD, Principal Investigator — University of Massachusetts, Worcester; Carol A Cicarrelli, RN, Study Director — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States